CLINICAL TRIAL: NCT01593020
Title: A Randomized Phase II Neoadjuvant Study of Sequential Eribulin Followed by FAC/FEC-regimen Compared to Sequential Paclitaxel Followed by FAC/FEC-Regimen in Women With Early Stage Breast Cancer Not Overexpressing HER-2
Brief Title: Neoadjuvant Study of Sequential Eribulin Followed by FAC Compared to Sequential Paclitaxel Followed by FEC in Early Stage Breast Cancer Not Overexpressing HER-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0167; NCI-2012-00851 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Early Stage Breast Cancer Not Overexpressing HER-2; Primary invasive adenocarcinoma of the breast; Paclitaxel; Taxol; Eribulin; E7389; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Epirubicin; Ellence; Cyclophosphamide; Cytoxan; Neosar; Doxorubicin; Doxorubicin hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; eribulin; Fluorouracil; Epirubicin; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paclitaxel + FEC or FAC Group (Experimental): ARM 1: Participants receive Paclitaxel 80 mg/m2 by vein over 1 hour weekly for 12 doses of a 21 day cycle.
  Participants on both arms receive FEC or FAC for 4 cycles (21 day cycle) at the preference of the treating physicians.
  Interventions: Drug: Paclitaxel; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Doxorubicin
- Eribulin + FEC or FAC Group (Experimental): ARM 2: Participants receive Eribulin 1.4 mg/m2 by vein over 2-5 minutes on days 1 and 8 every 3 weeks for 4 cycles (21 day cycle).
  Participants on both arms receive FEC or FAC for 4 cycles (21 day cycle) at the preference of the treating physicians.
  Interventions: Drug: Eribulin; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 by vein over 1 hour on Days 1, 8, and 15 of each 21-day cycle.
  Other Names: Taxol
  Arms: Paclitaxel + FEC or FAC Group
Drug: Eribulin — 1.4 mg/m2 by vein over 2-5 minutes on Days 1 and 8 of each 21-day study cycle.
  Other Names: E7389
  Arms: Eribulin + FEC or FAC Group
Drug: 5-Fluorouracil — 500 mg/m2 by vein on day 1 for 4 cycles (21 day cycle) at preference of treating physicians.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Epirubicin — 100 mg/m2 by vein on day 1 for 4 cycles (21 day cycle) at preference of treating physicians.
  Other Names: Ellence
Drug: Cyclophosphamide — 500 mg/m2 by vein on day 1 for 4 cycles (21 day cycle) at preference of treating physicians.
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 50 mg/m2 by vein on day 1, over 72 hour continuous infusion or intravenous bolus, for 4 cycles (21 day cycle) at preference of treating physicians.
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex

SUMMARY:
The goal of this clinical research study is to learn if and how well eribulin, given in combination with standard chemotherapy, can treat early-stage breast cancer compared to paclitaxel given in combination with standard chemotherapy. In this study, the standard chemotherapy being given is either 5-fluorouracil, epirubicin, and cyclophosphamide (called FEC) or 5-fluorouracil, doxorubicin, and cyclophosphamide (called FAC).

Eribulin is a changed version of the structure of a natural substance from a sea sponge. It is designed to block cells from dividing, which may cause cancer cells to die.

Paclitaxel is designed to block cancer cells from dividing, which may cause them to die.

5-fluorouracil is designed to block cancer cells from growing and dividing, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Epirubicin is designed to block the way cancer cells grow and divide, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Doxorubicin is designed to stop the growth of cancer cells, which may cause the cells to die.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and/or keep them from spreading throughout the body. This may cause the cancer cells to die.

DETAILED DESCRIPTION:
Study Groups If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to either group.

If you are in Group 1, you will receive paclitaxel for 4 cycles. You also will be treated with FAC or FEC for 4 cycles. Your treating doctor will decide whether you will receive FEC or FAC.

If you are in Group 2, you will receive eribulin for 4 cycles. You will also be treated with FAC or FEC for 4 cycles. Your treating doctor will decide whether you will receive FEC or FAC.

Each cycle is 21 days.

Study Drug Administration for Group 1 You will receive paclitaxel by vein over 1 hour on Days 1, 8, and 15 of each 21-day study cycle.

Before the infusion, you will be given drugs by vein, to help decrease the risk of an allergic reaction.

If you have severe side effects, future treatments may be delayed, the dose may be decreased, or you may be taken off study.

Once you have received 4 cycles of paclitaxel, you will receive either FEC or FAC chemotherapy for 4 cycles. Your treating doctor will decide whether you will receive FEC or FAC.

Study Drug Administration for Group 2 You will receive eribulin by vein over 2-5 minutes on Days 1 and 8 of each 21-day study cycle.

Once you have received 4 cycles of eribulin, you will receive FEC or FAC chemotherapy for 4 cycles. Your treating doctor will decide whether you will receive FEC or FAC.

FEC or FAC Treatment After you have received 4 cycles of either paclitaxel or eribulin, you will receive FEC or FAC.

If you are given FEC chemotherapy, you will receive 5-Fluorouracil by vein over 15 minutes, epirubicin by vein over 30 minutes, and cyclophosphamide by vein over 30-60 minutes on Day 1 of every 21-day cycle.

If you are given FAC chemotherapy, you will receive 5-Fluorouracil by vein over 15 minutes, doxorubicin by vein over 15 minutes, and cyclophosphamide by vein over 30-60 minutes on Day 1 of 21-day cycle.

Before FEC or FAC chemotherapy, you will be given drugs by vein to help decrease the risk of allergic reaction. These drugs will include dexamethasone and zofran.

Study Visits During Paclitaxel or Eribulin On Day 1 of each cycle: If you have had these tests within 10 days before Day 1 of Cycle 1, they may not need to be repeated.

You will have a physical exam, including a measurement of your weight and vital signs.

You will be asked about any side effects you may be having and any drugs you may be taking.

Your performance status will be recorded. Blood (about 1-2 teaspoons) will be drawn for routine tests.

On Days 8 and 15 of Cycle 1-4, blood (about 1 teaspoon) will be drawn for routine tests.

At Week 12, you will have a core biopsy.

At the end of Cycle 4:

You will have an ultrasound of the breast to check the status of the disease. You will have an ECHO or MUGA scan. You will have a core biopsy and fine needle aspiration of the tumor. A small needle will be inserted into the tumor at the safest and easiest location to withdraw cancer cells. This will be used to learn which tumor markers may predict who may best respond to therapy.

Study Visits During FEC or FAC Chemotherapy

On Day 1 of every third week:

You will have a physical exam, including a measurement of your weight and vital signs.

You will be asked about any side effects you may be having and any drugs you may be taking.

Your performance status will be recorded. Blood (about 1-2 teaspoons) will be drawn for routine tests.

After you have finished FEC or FAC treatment, you may have surgery. At the end of the chemotherapy treatment, you will be referred to the breast surgeon to discuss surgery. There is an small possibility (less than 3%) that tumor has gotten worse during treatment, and additional chemotherapy may be necessary.

Length of Study You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Paclitaxel, doxorubicin, epirubicin, and cyclophosphamide are FDA approved and commercially available for the treatment of breast cancer. Eribulin is FDA approved and commercially available to treat metastatic breast cancer in patients who have received at least 2 chemotherapy regimens for the treatment of metastatic disease. The use of eribulin with the FEC/FAC regimens is investigational for neoadjuvant treatment.

Eribulin will be provided at no cost to you while you are on this study. You and/or your insurance provider will be responsible for the cost of paclitaxel, doxorubicin, epirubicin, and cyclophosphamide.

Up to 162 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Histologically confirmed primary invasive adenocarcinoma of the breast.
3. Clinical stage breast cancer T2-3, N0-3, M0
4. Negative HER-2/neu expression as determined by local hospital laboratory using Fluorescence In Situ Hybridization (FISH), or is less or equal to 1+ using Immunohistochemistry (IHC).
5. No prior treatment for primary invasive adenocarcinoma of the breast such as irradiation, chemotherapy, hormonal therapy, immunotherapy, investigational therapy or surgery. Subjects receiving hormone replacement treatment (HRT) are eligible if this therapy is discontinued at least 2 weeks before starting study treatment. Treatment for DCIS is allowed, such as surgery, hormonal therapy and radiotherapy.
6. Karnofsky performance status (KPS) of 80 - 100
7. The ability and willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
8. Baseline MUGA or echocardiogram scans with LVEF of > 50%.
9. Normal PTT and either INR or PT < 1.5 x ULN.
10. Men or women 18 years of age or older.
11. Women of childbearing potential (WOCBP) must agree to use a medically acceptable method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of study drugs.
12. Willingness to have core biopsies and/or FNA performed before the start of study treatment and at the end of 12 week on treatment.

Exclusion Criteria:

1. Women who are pregnant (including positive pregnancy test at enrollment or prior to study drug administration) or breast-feeding.
2. Disease free of prior malignancy for < 5 years with the exception of DCIS, curatively treated basal carcinoma of the skin, local skin squamous cell carcinoma, or carcinoma in situ of the cervix.
3. Absolute neutrophils count (ANC) < 1500/mm^3
4. Total bilirubin > 1.5 times the upper limit of normal (ULN)
5. AST or ALT > 2.5 times the upper limit of normal (ULN)
6. Platelets < 100,000/mm^3.
7. Serum creatinine > 1.5 x ULN or creatinine clearance < 60 mL/min (measured or calculated by Cockcroft-Galt method)
8. Evidence of metastatic breast cancer following a standard tumor staging work-up
9. Evidence of inflammatory breast cancer.
10. Evidence of any grade 2 sensory or motor neuropathy.
11. Known human immunodeficiency viral (HIV) infection
12. Serious intercurrent infections or non-malignant medical illness that are uncontrolled or the control of which may be jeopardized by this therapy.
13. Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocols.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from August 2012 to July 2014. This study was conducted at the University of Texas MD Anderson Cancer Center main campus and the Regional Care Centers (RCC).
Pre-assignment Details: 54 patients were accrued. 28 patients were randomized to Paclitaxel and 26 patients to Eribulin group. 2 patients from eribulin were found ineligible and never received treatment and 1 patient withdrew due to physician decision.
Groups:
- Paclitaxel Weekly for 12 Doses Followed by FAC/FEC: Patients will receive Paclitaxel 80 mg/m2 IVPB over 1 hour weekly for 12 doses followed by FAC/FEC.
- Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC: Patients will receive eribulin 1.4 mg/m2 IV infusion or per institutional guidelines over 2-5 minutes on days 1 and 8 every 3 weeks for 4 cycles (21 day cycle) followed by FAC/FEC.
Period: Overall Study
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC
Started | 28 | 23
Completed | 26 | 21
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 20 | 48
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: Pathologic complete response (pCR) defined as complete absence of any viable invasive cancer cells in the resected breast and lymph nodes. Participants undergo definitive breast surgery 4 -6 weeks from last dose of FAC/FEC-regimen. Tumors removed by either lumpectomy with axillary dissection (i.e. breast conservation surgery) or modified radical mastectomy (i.e. mastectomy with axillary clearance). Surgical specimens (breast and axillary lymph node tissue) evaluated for pathological complete response.
Time Frame: 4 -6 weeks from last dose of FAC/FEC-regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC
Number analyzed (Participants) | 26 | 21
Participants | 7 | 1

2. Secondary Outcome: 5 Year Event Free Survival (EFS)
Description: Event free survival (EFS) the length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Time Frame: from start of treatment, up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC
Number analyzed (Participants) | 28 | 23
percentage of participants | 81.8 | 74

3. Secondary Outcome: Overall Survival (OS)
Time Frame: from start of treatment, up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC
Number analyzed (Participants) | 28 | 23
percentage of participants | 100 | 84.4

ADVERSE EVENTS:
Time Frame: The duration of chemotherapy treatment per subject will be approximately 6 months, corresponding to 4 cycles of eribulin followed by 4 cycles of FAC/FEC-regimen or 12 cycles of weekly paclitaxel followed by 4 cycles of FAC/FEC-regimen. Post chemotherapy, patient will undergo definitive breast surgery 4 -6 weeks from last dose of FAC/FEC-regimen. 2 weeks Follow up post surgery
Description: Only >/= grade 3 serious adverse events are reported
Arm/Group | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/23
Serious Adverse Events (participants affected / at risk) | 3/28 | 9/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Weekly for 12 Doses Followed by FAC/FEC (N=28) | Eribulin on Days 1 and 8 Every 3 Weeks for 4 Cycles (21 Day Cycle) Followed by FAC/FEC (N=23)
Fatigue (General disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (3) | 9 (9)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT01593020/Prot_SAP_000.pdf